CLINICAL TRIAL: NCT03544736
Title: Safety and Feasibility of Irradiation and Nivolumab in Esophageal Cancer (INEC-study) - a Phase I/II Trial
Brief Title: Safety and Feasibility of Irradiation and Nivolumab in Esophageal Cancer (INEC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Geir Olav Hjortland, Principal Investigator, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9M9-03
Record Dates: First submitted 2018-04-25; First posted 2018-06-04 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Cancer
Keywords: Nivolumab; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nivolumab; Radiotherapy; Drug Therapy; Paclitaxel; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, Parallell Groups, Study of Nivolumab and Radiotherapy in Patients With Esophageal Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Subjects having palliative radiotherapy towards esophageal tumor will receive concomitant therapy With Nivolumab i.v. 240mg Q2W: first 6 patients, 360mg Q3W: Next 6 patients or 480mg Q4W: Last 6 patients, treatment to progression or up to 2 years of treatment.
  Radiotherapy: 2 Gy / day, (5 fx/week) to a total of 20 - 50 Gy in 25fx (2-4Gy/fx) at the decision of the responsible physician.
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy
- Cohort B (Experimental): Subjects receiving definitive chemoradiotherapy for esophageal cancer will receive concomitant therapy with Nivolumab 240mg Q2W, during RT, and continued with 480mg Q4W, treatment to progression or up to 1 year after completion of radiotherapy. 6 patients in total.
  Chemotherapy: Paclitaxel i.v. 175mg/m2 and Carboplatin AUC5, then after 21 days Radiotherapy 1,8 Gy / day (5 fx/week) up to 50,4 Gy in 28fx and concomitantly Paclitaxel 50mg/m2 and Carboplatin AUC2 Q1W and Nivolumab as described above.
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy; Drug: Chemotherapy
- Cohort C (Experimental): Subjects with operable esophageal cancer eligible for neoadjuvant chemoradiotherapy will receive Nivolumab 240mg Q2W, concomitantly with RT Then surgery 4-12 weeks after RT. Within 6-12 months after surgery: Adjuvant Nivolumab 480mg Q4W, for 12 months. 6 patients in total.
  Neoadjuvant chemotherapy: Concomitantly Paclitaxel 50mg/m2 and Carboplatin AUC2 Q1W and Radiotherapy: 41,4 Gy in 23 fractions.
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy; Drug: Chemotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Nivolumab — Experimental: Nivolumab
  Other Names: Opdivo
Radiation: Radiotherapy — Radiotherapy
Drug: Chemotherapy — Chemotherapy
  Other Names: Paclitaxel and Carboplatin
  Arms: Cohort B; Cohort C
Procedure: Surgery — Surgery
  Arms: Cohort C

SUMMARY:
Three parallel cohort, multicenter, open-label, phase I/II clinical trial to analyze the safety and feasibility of PD-1 inhibition with Nivolumab given concomitantly with standard radiotherapy regimens in the treatment of esophageal cancer

DETAILED DESCRIPTION:
Three parallel cohort, multicenter, open-label, phase I/II clinical trial to analyze the safety and feasibility of PD-1 inhibition with Nivolumab given concomitantly with standard radiotherapy regimens in the treatment of esophageal cancer.

Cohort A: Advanced/inoperable esophageal cancer, eligible for palliative radiotherapy of the primary tumor.

Cohort B: Inoperable esophageal cancer without metastases, eligible for definitive chemoradiotherapy Cohort C: Operable esophageal cancer eligible for neoadjuvant chemoradiotherapy

ELIGIBILITY:
Inclusion Criteria:

Three different cohorts of patients with esophageal cancer are studied.

All of the following conditions must apply to the prospective patient at screening prior to receiving study treatment or any study related procedures (e.g.):

* Age > 18 years
* Patients should have previously untreated histologically proven squamous cell carcinoma or adenocarcinoma of the esophagus or the gastroesophageal junction (GEJ), Siewert I, II or III
* Must be ambulatory with a performance status ECOG 0 or 1
* Adequate organ function based on clinical examination and lab values as defined in the below:

Absolute neutrophil count: ≥ 1,5 x109/L Platelets: ≥ 100 x109/L Hemoglobin: ≥ 9 x109/L Creatinine ≤ 1,5 upper limit normal (ULN) OR measured/calculated GFR≥60 mL/min Albumin ≥ 30 g/L Total bilirubin ≤ 1,5 ULN ASAT and ALAT ≤ 2,5 ULN, or ≤ 5 ULN for subjects with liver mets. International Normalized Ratio (INR) ≤ 1,5 ULN and Activated Partial Thromboplastin Time (TT) ≤ 1,5 ULN unless subject is receiving anticoagulant therapy. Such therapy (if indicated) should be converted to adequate therapy with low-molecular weight heparin such as Dalteparin before chemotherapy or treatment with IMP.

* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 28 days prior to the start of study drug (screening phase). Women must not be breastfeeding.
* WOCBP should use highly effective adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of investigational drug. Adequate methods are described in Appendix I.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception during the study treatment period and until 7 months after last dose of Nivolumab (see Appendix I).
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.
* If Dysphagia score >2, a nasogastric feeding tube should be inserted during the aid of gastroscopy, and nasogastric tube feeding started before radiotherapy.
* In addition, specific criteria are defined for the three different patient cohorts below:

Specific inclusion criteria - Cohort A

* Eligible for palliative fractionated radiotherapy of the esophageal- or gastroesophageal cancer as determined by the multidisciplinary team (MDT) meeting.
* Expected survival >3 months
* Not bulky disease, i.e. palliative radiotherapy towards the primary tumor is intended to palliate dysphagia and/or pain and systemic treatment could be delayed to AFTER protocol therapy if possible.

Specific inclusion criteria - Cohort B

* Eligible for definitive chemoradiation of localized but inoperable esophageal- or gastroesophageal cancer as determined by the multidisciplinary team (MDT) meeting.
* Regional disease, i.e. no metastasis outside the radiation field (PTV).
* Considered candidate/ able to adhere to the intended chemoradiotherapy

Specific inclusion criteria - Cohort C

* Eligible for neoadjuvant chemoradiotherapy and surgery of the esophageal- or gastroesophageal cancer as determined by the multidisciplinary team (MDT) meeting.
* Regional disease, i.e. no metastasis outside the radiation field (PTV).
* Considered candidate and able to adhere to the intended neoadjuvant chemoradiotherapy and planned surgery.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Previous treatment with radiotherapy towards volumes within the thoracic cavity
* Previous treatment with any PD-1 or PD-L1/2 inhibitor
* Hypersensitivity to the investigational product or any of the drug formula contents
* Esophageal stenting
* T4b if infiltration into the aorta or the trachea
* History of prior autoimmune disorders requiring systemic therapy (excluding Insulin or Thyroid replacement therapy)
* History of HIV 1 /2, Hepatitis B or C infection
* History of Immunodeficiency disorders (i.e. immunoglobulin deficiency or white blood cell lineage depletion disorders)
* Participation in any other interventional clinical trial with an investigational product
* History of prior malignancy within the last 5 years, excluding curatively treated basal cell or squamous cell carcinoma of the skin.
* Known history of brain metastases
* Need to use immunosuppressive drugs including, but not limited to: Glucocorticoids, everolimus, sirolimus, disease-modifying anti-rheumatic drugs (DMARDS)
* Positive pregnancy test (positive hCG blood test)
* Known allergy, hypersensitivity, or contraindication to the investigational product Nivolumab, or the drugs paclitaxel and docetaxel used in the standard chemoradiotherapy protocols (Cohorts B and C) or any components used in their preparation or has a contraindication to taxane therapy.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of treatment allocation until first date of documented disease progression or death assessed during study period or up to at least 100 days after last dose
  Safety and Tolerability; Incidence of adverse events using CTCAE 5.0

SECONDARY OUTCOMES:
Response to treatment | From date of treatment allocation and during treatment period up to 2 years
  Overall Response Rate (RECIST v1.1)
Overall Survival | From date of treatment allocation until first date of documented death assessed up to 5 years after completed treatment
  The survival time from date of treatment allocation until first date of documented death
Progression Free Survival | From date of treatment allocation until first date of documented disease progression or death assessed up to 5 years after completed treatment
  The time from date of treatment allocation until first date of documented disease progression or death whichever comes first
Health Related Quality of Life (EQ-5D) | From date of treatment allocation until first date of documented disease progression or death assessed up to 5 years after completed treatment
  Health Related Quality of Life Measurements, using patients' reported outcomes from EQ-5D
Health Related Quality of Life (EORTC QLQ-C30) | From date of treatment allocation until first date of documented disease progression or death assessed up to 5 years after completed treatment
  Health Related Quality of Life Measurements, using patients' reported outcomes from EORTC QLQ-C30
Health Related Quality of Life (EORTC QLQ-OG25) | From date of treatment allocation until first date of documented disease progression or death assessed up to 5 years after completed treatment
  Health Related Quality of Life Measurements, using patients' reported outcomes from EORTC QLQ-OG25

CONTACTS AND LOCATIONS:
Overall Officials: Geir O. Hjortland, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway